CLINICAL TRIAL: NCT04584424
Title: Prognostic Factors and Outcomes of COVID-19 Cases in Ethiopia: Multi-Site Cohort Study
Brief Title: Prognostic Factors and Outcomes of COVID-19 Cases in Ethiopia
Status: Completed | Type: Observational
Sponsor: Ethiopian Public Health Institute (Other Government)
Responsible Party: Principal Investigator, Masresha Tessema, Principal Investigator, Ethiopian Public Health Institute
Other Study IDs: EPHI National Cohort
Record Dates: First submitted 2020-09-22; First posted 2020-10-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Epidemiology; Clinical; Nutritional-status; Immunologic Defect
Keywords: Ethiopia, Epidemiological and Clinical features of COVID-19 cases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — i. Laboratory diagnosis of SARS-CoV-2 infection: Patients' nasopharyngeal/through swab specimens will be collected for the SARS-CoV-2 viral nucleic acid detection using real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay.
  ii. Phylogenetic analysis of SARS-CoV-2. iii. Imaging: Chest x-ray, chest computed tomographic (CT) scans data will be retrieved if available.
  iv. Clinical chemistry: Albumin, Fibrinogen level, lactate dehydrogenase, alanine aminotransferase, aspartate aminotransferase, total bilirubin, creatinine, cardiac troponin, D-Dimer, pro-calcitonin and C-reactive protein, and vitamin D concentration will be assessed using fully automated Cobas 6000.
  v. Serum levels of Anti-SARS-CoV-2 IgM, IgG or IgM/IgG antibodies, selected pro-inflammatory cytokines, anti-inflammatory or regulatory cytokines and chemokines will be measured using rapid or ELISA based platforms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The study does not required — The study is prospective multi-center COVID-19 patient cohort

SUMMARY:
The aim of the study will be to determine the epidemiological and clinical features of COVID-19 cases, immunological and virological courses, interaction with nutritional status, and response to treatment for COVID-19 patients admitted to treatment centers in Ethiopia.

Methods: This multi-site cohort enrolls, patients with confirmed COVID-19 infection admitted to treatment centers will be enrolled irrespective of their symptoms and followed up for 12 months. Baseline epidemiological, clinical, laboratory and imaging data will be collected from treatment records, interviews, physical measurements and biological samples. Endline data involves treatment and prognostic outcomes to be measured using different biomarkers and clinical parameters, The patients will be followed up in the selected treatment centers for COVID-19 infection. For all data collected both descriptive and multivariable analyses will be performed to isolated determinants of the treatment outcome and prognosis to generate relevant information for informed prevention and case management.

DETAILED DESCRIPTION:
Background: The coronavirus disease 2019 (COVID-19) became pandemic after emerging in Wuhan, China, in December 2019 which is caused by severe acute respiratory syndrome coronavirus (SARS-CoV-2). Following the swift spread of the virus,4, 710,000 confirmed cases and 315,000 deaths were reported worldwide as of May 17, 2020,and 317 confirmed cases and 5 deaths are reported nationally. To understand the drastically negative impacts of COVID-19 on the public health and key features pertinent to the disease various researches are under investigation at the global level and they are contributing to delineating the characteristics of the disease and its lethality. However, the potential acceptability of different risks varies depending on numerous factors including the type of research and the context in which it takes place. Currently, it is recognized that a 'one size fits all' approach towards the design and implementation of interventions may not be appropriate. Therefore, it is found apparent that global priorities, protocols and intervention assessments have to be contextualized and adjusted to local needs and realities, including translation of results.

Objective: To determine the epidemiological and clinical features of COVID-19 cases, immunological and virological courses, interaction with nutritional status, and response to treatment for COVID-19 patients admitted to treatment centers in Ethiopia.

Methods: This multi-site cohort enrolls, patients with confirmed COVID-19 infection admitted to treatment centers will be enrolled irrespective of their symptoms and followed up for 12 months. Baseline epidemiological, clinical, laboratory and imaging data will be collected from treatment records, interviews, physical measurements and biological samples. Endline data involves treatment and prognostic outcomes to be measured using different biomarkers and clinical parameters, The patients will be followed up in the selected treatment centers for COVID-19 infection. For all data collected both descriptive and multivariable analyses will be performed to isolated determinants of the treatment outcome and prognosis to generate relevant information for informed prevention and case management.

Expected outcome: The study will generate scientific data for a systematic understanding of natural history, epidemiological characteristics, clinical features and management of COVID-19 that will in turn enables country's health sector to develop strategies to prevent and control the pandemic before it poses further health and socioeconomic crisis.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to treatment centers, with confirmed SARS-CoV-2 infection (virologically confirmed diagnosis by RT-PCR).
* Agrees to be enrolled in the follow-up study and provide all necessary information/data, blood and nasopharyngeal swab for testing.

Exclusion Criteria:

* A subject deprived of freedom, subject under a legal protective measure
* Refusal by participant, parent or appropriate guardian or representative
* Confirmed diagnosis of other pathogens unrelated to the objectives of this study and no indication or likelihood of co-infection with a relevant pathogen.
* Participants who will not willing to stay 12 months in the cohort in Ethiopia.
* Those who are prior involved in the COVID-19 clinical trial or other intervention studies.
* Not capable of understanding or complying with the study protocol or provide consent
* Anticipated transfer to another hospital that is not a study site within 72 hours
* Patients who cannot stand straight due to amputation, kyphosis, scoliosis or paralyzes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be confirmed SARS-CoV-2 infection (virologically confirmed diagnosis by RT-PCR). This will include both symptomatic (sever, moderate and critical cases) and asymptomatic patients.
Sampling Method: Probability Sample
Enrollment: 6390 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Number of patients survival or death | 12 months
  Number patients developing severe infection or death
Rate of recovery time | 4 weeks
  Mean rate of recovery in patients with diagnosis of COVID-19
Viral shedding | 6 weeks
  proportion of shedding detected in environment and personal protective equipment

SECONDARY OUTCOMES:
Viral loads | 12 months
  quantity of viral load
Clinical symptoms and signs | 12 months
  clinical manifestations Proportions of mild, moderate, severe and critical cases
Blood pressure | 4 weeks
  Force exerted by the blood against the walls of the vessels (arteries) as it is pumped by the heart. Measurement using the multi-parameter vital signs monitor. Units of measurement in mmHg. Obtain systolic and diastolic pressure.
Assess the prevalence of severe forms among hospitalized patients with diabètes and COVID-19 | 4 weeks
  Prevalence of severe forms among all COVID-19 patients with diabetes
Assess the prevalence of severe forms among hospitalized patients with cancer and COVID-19 | 4 weeks
  proportion of patients with cancer and COVID-19 postive
Lipid Profiles | 12 months
  TC, TG, HDL-C, and LDL-C
Assess the prevalence of nutrient intakes | 12 months
  Prevalence of inadequate intake of zinc, Iron and Vitamin A
Assess the prevalence of micronutrients deficiencies among hospitalized patients with COVID-19 | 12 months
  Prevalence of Vitamin D, zinc, and Iron deficiency anemia measured in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Saro Abdella, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The di-identified datasets after reaching objectives of the study could shared. Interested researchers can request investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available upon compilation of the data collection and cleaning
Access Criteria: This may depend on the request and objectives.

REFERENCES:
- [Derived] Abdella S, Tessema M, Tasew G, Defar A, Deressa A, Regasa F, Teka F, Tigabu E, Nigussie D, Belachew T, Molla M, Deribew A, Abebe W, Yigzaw T, Nigatu T, Mitike G, Haile T, Taame H, Ahmed M, Nigatu F, Tolesa T, Wolka E, Amogne W, Laillou A, Amare M, Fufa Y, Argaw A, Waganew W, Azazh A, Worku A, Redae B, Sultan M, Walelegn M, Tefera M, Yifru S, Argaw R, Brehau N, Teklu S, Demoz G, Seman Y, Salasibew M, Ejeta E, Whiting SJ, Wolday D, Tollera G, Abate E, Duguma D. Prognostic factors and outcomes of COVID-19 cases in Ethiopia: multi-center cohort study protocol. BMC Infect Dis. 2021 Sep 16;21(1):956. doi: 10.1186/s12879-021-06652-0. PMID 34530744